CLINICAL TRIAL: NCT00401960
Title: Open Label Study to Assess the Efficacy and Safety of Daptomycin in Combination With Anti-Cell Wall Active Therapy in the Treatment of Enterococcal Endocarditis
Brief Title: Daptomycin as an Adjuvant Agent in the Treatment of Enterococcal Native Valve Endocarditis.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: inadequate enrollment
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Rhee, Kyu Y., Assistant Professor, Weill Medical College of Cornell University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0507008023
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Endocarditis, Bacterial
Keywords: Enterococcus; Daptomycin; Endocarditis
MeSH Terms: conditions — Endocarditis, Bacterial; Endocarditis | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daptomycin adjunctive group (Experimental): Patients with enterococcal endocarditis who elect to receive daptomycin at a dose of 8 milligrams/kilogram/day in addition to the antibiotics they are already receiving
  Interventions: Drug: Daptomycin
- standard of care (No Intervention): Patients with enterococcal endocarditis who elect to receive standard of care therapy as prescribed by their primary physician

INTERVENTIONS:
Drug: Daptomycin — daptomycin at a dose of 8 milligrams/kilogram/day in addition to the antibiotics they are already receiving for native valve enterococcal endocarditis
  Other Names: Cubicin
  Arms: Daptomycin adjunctive group

SUMMARY:
The aim of this study is to determine the safety and efficacy of daptomycin when used as an adjuvant agent to standard care in the treatment of proven native valve Enterococcal endocarditis. Patients with this disease will be offered the option of receiving daptomycin at a dose of 8 milligrams/kilogram/day in addition to the antibiotics they are already receiving. The hypothesis of this study is that daptomycin added to standard therapy for Enterococcal endocarditis is safe and efficacious.

Patients who receive daptomycin + standard therapy will be compared to patients who receive standard therapy alone with respect to the following outcomes:

1. Safety.

   1. The frequency of any Grade 3 or 4 toxicity (DAIDS scale) will be measured.
   2. The frequency of muscle toxicity or renal toxicity, as determined by predefined criteria.
2. Efficacy.

   1. Clinical efficacy.

      * Time to clearance of bacteremia
      * Cure at 6 weeks following completion of antibiotic therapy
      * Mortality at 6 weeks following completion of antibiotic therapy
   2. Microbiologic efficacy.

      * Peak and trough serum bactericidal titers
      * The minimum bactericidal concentration of Enterococci to daptomycin

We expect to enroll 40 patients over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Definite Enterococcal endocarditis, as defined by modified Duke criteria
* Able to complete follow-up 3 and 6 weeks following completion of intravenous antibiotic therapy

Exclusion Criteria:

* Pregnancy or breast feeding
* Creatine phosphokinase levels over two times the upper limit of normal
* Renal insufficiency or dialysis requirement.
* Presence of chronic indwelling bloodstream catheters or foreign body devices suspected as primary or secondary sites of enterococcal infection unamenable to removal or replacement
* Inability to discontinue or abstain from use of a HMG CoA reductase inhibitor during the study period.
* Hypersensitivity to any of the study medications.
* Any condition that, in the investigator's opinion, may interfere with protocol compliance including, but not limited to, active substance abuse and/or dementia.
* Prosthetic valve endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Y Rhee, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NewYork-Presbyterian Hospital, Weill Cornell Campus, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This was a pilot single arm study, for which IPD are not pertinent

RESULTS

PARTICIPANT FLOW:
Groups:
- Adjunctive Daptomycin Group: please see study description for study enrollment
- Standard of Care Group: as per study description
Period: Overall Study
Arm/Group | Adjunctive Daptomycin Group | Standard of Care Group
Started | 5 | 1
Completed | 0 | 1
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Population: see study inclusion criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjunctive Daptomycin Group | Standard of Care Group | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 69 [31 to 88] | 74 [74 to 74] | 70 [31 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Grade 3 or 4 Toxicity (DAIDS Scale)
Description: Number of Participants any Grade 3 or 4 toxicity (DAIDS scale); please see adverse event table for details
Time Frame: weekly
Population: Study terminated due to insufficient enrollment; therefore data not sufficient for planned analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Adjunctive Daptomycin Group | Standard of Care Group
Number analyzed (Participants) | 5 | 1
Participants | 4 | 0

2. Primary Outcome: Number of Participants With Muscle Toxicity or Renal Toxicity, as Determined by Predefined Criteria
Description: Number of Participants with creatine kinase elevation > 3x upper limit of normal or elevations of serum Cr >= 30% above baseline
Time Frame: weekly
Population: study terminated due to inadequate enrollment; therefore data not sufficient for planned analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Daptomycin Adjunctive Group | Standard of Care
Number analyzed (Participants) | 5 | 1
Participants
  Elevated serum creatinine >= 30% above baseline | 1 | 1
  Elevate serum creatine kinase > 3X ULN | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years; however, study terminated due to lack of eligible study participants
Arm/Group | Adjunctive Daptomycin Group | Standard of Care Group
Serious Adverse Events (participants affected / at risk) | 5/5 | 0/1
Other Adverse Events (participants affected / at risk) | 0/5 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjunctive Daptomycin Group (N=5) | Standard of Care Group (N=1)
hemopericardium (Cardiac disorders) | 2 (2) | 0 (0) — underlying rheumatic heart disease and congestive heart failure; underlying conduction disorder S/P pacemekaer; both deemed unrelated to antibiotics
death (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — uncontrolled progression of underlying CLL
Cr elevation (Renal and urinary disorders) | 1 (1) | 0 (0) — day 9 of combination ABX with ampicillin, gentamicin, daptomycin- possibly related to daptomycin
death (Infections and infestations) | 1 (1) | 0 (0) — nosocomial Serratia pneumonia

LIMITATIONS AND CAVEATS:
study terminated due to insufficient enrollment; data therefore not analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No